CLINICAL TRIAL: NCT00788541
Title: A Dose-Volume Study of the Safety and IOP-Lowering Efficacy of Anecortave Acetate in Patients With Open-Angle Glaucoma or Ocular Hypertension
Brief Title: A Dose-Volume Study of a Treatment for Elevated IOP Due to Open-Angle Glaucoma or Ocular Hypertension
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Project cancellation
Sponsor: Alcon Research (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: C-08-049
Record Dates: First submitted 2008-11-07; First posted 2008-11-11 (Estimated); Last update posted 2012-11-30 (Estimated); Status verified 2012-11

CONDITIONS: Open-Angle Glaucoma; Ocular Hypertension
Keywords: Open-Angle Glaucoma; Intraocular Pressure; Anecortave Acetate
MeSH Terms: conditions — Glaucoma, Open-Angle; Ocular Hypertension | interventions — anecortave acetate

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (6):
- 3 mg Anecortave Acetate, low volume high dose (Experimental): Anecortave Acetate Sterile Suspension, 6 mg/mL, one injection of 0.5 mL in the study eye monthly for 6 months.
  Interventions: Drug: Anecortave Acetate Sterile Suspension, 6 mg/mL
- 3 mg Anecortave Acetate, high volume low dose (Experimental): Anecortave Acetate Sterile Suspension, 3.75 mg/mL, one injection of 0.8 mL in the study eye monthly for 6 months.
  Interventions: Drug: Anecortave Acetate Sterile Suspension, 3.75 mg/mL
- 48 mg Anecortave Acetate, low volume high dose (Experimental): Anecortave Acetate Sterile Suspension, 96 mg/mL, one injection of 0.5 mL in the study eye monthly for 6 months.
  Interventions: Drug: Anecortave Acetate Sterile Suspension, 96 mg/mL
- 48 mg Anecortave Acetate, high volume low dose (Experimental): Anecortave Acetate Sterile Suspension, 60 mg/mL, one injection of 0.8 mL in the study eye monthly for 6 months.
  Interventions: Drug: Anecortave Acetate Sterile Suspension, 60 mg/ML
- Anecortave Acetate Vehicle, low volume (Placebo Comparator): Anecortave Acetate Vehicle, one injection of 0.5 mL in the study eye monthly for 6 months.
  Interventions: Other: Anecortave Acetate Vehicle
- Anecortave Acetate Vehicle, high volume (Placebo Comparator): Anecortave Acetate Vehicle, one injection of 0.8 mL in the study eye monthly for 6 months.
  Interventions: Other: Anecortave Acetate Vehicle

INTERVENTIONS:
Drug: Anecortave Acetate Sterile Suspension, 6 mg/mL — Administered as an injection into an anterior juxtascleral depot
  Arms: 3 mg Anecortave Acetate, low volume high dose
Drug: Anecortave Acetate Sterile Suspension, 3.75 mg/mL — Administered as an injection into an anterior juxtascleral depot
  Arms: 3 mg Anecortave Acetate, high volume low dose
Drug: Anecortave Acetate Sterile Suspension, 96 mg/mL — Administered as an injection into an anterior juxtascleral depot
  Arms: 48 mg Anecortave Acetate, low volume high dose
Drug: Anecortave Acetate Sterile Suspension, 60 mg/ML — Administered as an injection into an anterior juxtascleral depot
  Arms: 48 mg Anecortave Acetate, high volume low dose
Other: Anecortave Acetate Vehicle — Administered as an injection into an anterior juxtascleral depot
  Arms: Anecortave Acetate Vehicle, high volume; Anecortave Acetate Vehicle, low volume

SUMMARY:
The purpose of this study was to assess the effects of total volume and total dose on the safety and intraocular pressure-lowering efficacy of Anecortave Acetate Suspension (3 mg and 48 mg) in 0.5 mL and 0.8 mL volumes when administered by anterior juxtascleral depot (AJD) for the treatment of elevated intraocular pressure (IOP) in patients with open-angle glaucoma or ocular hypertension.

ELIGIBILITY:
Inclusion Criteria:

* Clinical diagnosis of Open-Angle Glaucoma or Ocular Hypertension for at least 6 months;
* Other protocol-defined inclusion criteria may apply.

Exclusion Criteria:

* Prior angle surgery in the study eye, severe visual field loss in either eye;
* Other protocol-defined exclusion criteria may apply.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 197 (Actual)
Dates: Start 2008-12; Primary Completion 2009-09 (Actual); Study Completion 2009-09 (Actual)

PRIMARY OUTCOMES:
Mean Intraocular Pressure | 6 months

SECONDARY OUTCOMES:
Percent of patients who remain rescue-medication free | 6 Months

CONTACTS AND LOCATIONS:
Locations (1):
- Contact Alcon Call Center For Trial Locations, Fort Worth, Texas, United States